CLINICAL TRIAL: NCT04913337
Title: A Phase 1/2 Dose Escalation/Expansion Study of NGM707 As Monotherapy and in Combination with Pembrolizumab in Advanced or Metastatic Solid Tumor Malignancies
Brief Title: Study of NGM707 As Monotherapy and in Combination with Pembrolizumab in Advanced or Metastatic Solid Tumor Malignancies
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NGM Biopharmaceuticals, Inc (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 707-IO-101; KEYNOTE-D25 (Other: Merck Sharp & Dohme Corp); MK-3475-D25 (Other: Merck Sharp & Dohme Corp)
Record Dates: First submitted 2021-05-20; First posted 2021-06-04 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-06

CONDITIONS: Mesothelioma; Glioblastoma; Renal Cell Carcinoma; Non Small Cell Lung Cancer; Melanoma; Pancreatic Ductal Adenocarcinoma; Gastric Cancer; Squamous Cell Carcinoma of Head and Neck; Cholangiocarcinoma; Breast Cancer; Ovarian Cancer; Cervical Cancer; Endocervical Cancer; Colorectal Cancer; Esophageal Cancer
MeSH Terms: conditions — Mesothelioma; Glioblastoma; Carcinoma, Renal Cell; Carcinoma, Non-Small-Cell Lung; Melanoma; Stomach Neoplasms; Squamous Cell Carcinoma of Head and Neck; Cholangiocarcinoma; Breast Neoplasms; Ovarian Neoplasms; Uterine Cervical Neoplasms; Colorectal Neoplasms; Esophageal Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- NGM707 Monotherapy Dose Escalation (Experimental): Part 1a Single Agent Dose Escalation
  Interventions: Drug: NGM707
- NGM707 Combination Dose Finding with pembrolizumab (KEYTRUDA®) (Experimental): Part 1b NGM707 plus pembrolizumab (KEYTRUDA®)
  Interventions: Drug: NGM707 plus pembrolizumab (KEYTRUDA®)
- NGM707 Combination Dose Expansion Arm A (Experimental): NGM707 with pembrolizumab (KEYTRUDA®) in Squamous NSCLC
  Interventions: Drug: NGM707 plus pembrolizumab (KEYTRUDA®)
- NGM707 Combination Dose Expansion Arm B (Experimental): NGM707 with pembrolizumab (KEYTRUDA®) in Non-Squamous NSCLC
  Interventions: Drug: NGM707 plus pembrolizumab (KEYTRUDA®)
- NGM707 Combination Dose Expansion Arm C (Experimental): NGM707 with pembrolizumab (KEYTRUDA®) in SCCHN
  Interventions: Drug: NGM707 plus pembrolizumab (KEYTRUDA®)
- NGM707 Monotherapy Dose Expansion Arm D (Experimental): NGM707 in RCC
  Interventions: Drug: NGM707
- NGM707 Monotherapy Dose Expansion Arm E (Experimental): NGM707 in CRC
  Interventions: Drug: NGM707
- NGM707 Monotherapy Dose Expansion Arm F (Experimental): NGM707 in Ovarian
  Interventions: Drug: NGM707

INTERVENTIONS:
Drug: NGM707 — Drug: NGM707
  NGM707 is given intravenously (IV) every 3 weeks in a 21 day cycle. Multiple dose levels will be evaluated.
  Arms: NGM707 Monotherapy Dose Escalation
Drug: NGM707 plus pembrolizumab (KEYTRUDA®) — Drug: NGM707
  NGM707 is given intravenously (IV) every 3 weeks in a 21 day cycle. Multiple dose levels will be evaluated.
  Drug: pembrolizumab (KEYTRUDA®)
  Pembrolizumab (KEYTRUDA®) will be administered intravenously (IV) every 3 weeks in a 21 day cycle.
  Arms: NGM707 Combination Dose Finding with pembrolizumab (KEYTRUDA®)
Drug: NGM707 plus pembrolizumab (KEYTRUDA®) — Drug: NGM707
  NGM707 is given intravenously (IV) every 3 weeks in a 21 day cycle. Multiple dose levels will be evaluated.
  Drug: pembrolizumab (KEYTRUDA®)
  Pembrolizumab (KEYTRUDA®) will be administered intravenously (IV) every 3 weeks in a 21 day cycle.
  Arms: NGM707 Combination Dose Expansion Arm A
Drug: NGM707 plus pembrolizumab (KEYTRUDA®) — Drug: NGM707
  NGM707 is given intravenously (IV) every 3 weeks in a 21 day cycle. Multiple dose levels will be evaluated.
  Drug: pembrolizumab (KEYTRUDA®)
  Pembrolizumab (KEYTRUDA®) will be administered intravenously (IV) every 3 weeks in a 21 day cycle.
  Arms: NGM707 Combination Dose Expansion Arm B
Drug: NGM707 plus pembrolizumab (KEYTRUDA®) — Drug: NGM707
  NGM707 is given intravenously (IV) every 3 weeks in a 21 day cycle. Multiple dose levels will be evaluated.
  Drug: pembrolizumab (KEYTRUDA®)
  Pembrolizumab (KEYTRUDA®) will be administered intravenously (IV) every 3 weeks in a 21 day cycle.
  Arms: NGM707 Combination Dose Expansion Arm C
Drug: NGM707 — Drug: NGM707
  NGM707 is given intravenously (IV) every 3 weeks in a 21 day cycle. Multiple dose levels will be evaluated.
  Arms: NGM707 Monotherapy Dose Expansion Arm D
Drug: NGM707 — Drug: NGM707
  NGM707 is given intravenously (IV) every 3 weeks in a 21 day cycle. Multiple dose levels will be evaluated.
  Arms: NGM707 Monotherapy Dose Expansion Arm E
Drug: NGM707 — Drug: NGM707
  NGM707 is given intravenously (IV) every 3 weeks in a 21 day cycle. Multiple dose levels will be evaluated.
  Arms: NGM707 Monotherapy Dose Expansion Arm F

SUMMARY:
Study of NGM707 as Monotherapy and in Combination with Pembrolizumab in Advanced or Metastatic Solid Tumor Malignancies

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented locally advanced or metastatic solid tumor malignancy.
* Progressed or was intolerant to all available therapies known to confer clinical benefit appropriate for their tumor type, and for which the patient was eligible and willing to receive, or refused SOC treatments that are perceived to have marginal clinical benefit.
* Adequate bone marrow, kidney and liver function.
* Performance status of 0 or 1.
* Resolved acute effects of any prior therapy to baseline severity or CTCAE Grade 1 except for AEs not constituting a safety risk by Investigator judgement.

Exclusion Criteria:

* Prior treatment targeting ILT2 and/or ILT4 or targeting HLA-G.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Estimated)
Dates: Start 2021-06-09 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Dose-limiting Toxicities | Baseline up to 28 Days
  A DLT is defined as an AE that meets at least one of the criteria listed in protocol, according to National Cancer Institute (NCI) common terminology criteria for AE (CTCAE) version 5.0, and is considered by the investigator to be clinically relevant and attributed to the study treatment during the first 28 days after the first dose of study treatment.
Incidence of Adverse Events | Baseline up to Approximately 24 Months
  Number of patients with adverse events (AEs) according to severity, seriousness, and relationship to study drug
  An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of patients who experience at least one AE will be presented.
Number of Patients with Clinically Significant Laboratory Abnormalities | Baseline up to Approximately 24 Months
  Number of patients with clinically significant change from baseline in laboratory abnormalities as characterized by type, frequency, severity (graded by CTCAE version 5.0) and timing.
Number of Patients in Expansion Cohorts with Objective Responses | Baseline up to approximately 24 months
  Objective Response Rate is defined as the proportion of patients who achieve a confirmed complete response (CR) or partial response (PR) according to RECIST v1.1
Duration of Response for Patients in Expansion Cohorts | Baseline up to approximately 24 months
  Duration of Response is defined as the time from the first documentation of objective response (CR or PR) that is subsequently confirmed per RECIST v1.1, to the time of the first documentation of objective tumor progression or to death due to any cause, whichever occurs first.
Progression-free Survival for Patients in Expansion Cohorts | Baseline up to approximately 24 months
  Progression-free survival is defined as the time from start of study treatment to the date of first documentation of objective tumor progression on or following study therapy per RECIST v1.1, or to death due to any cause, whichever comes first.
Overall Survival for Patients in Combination Dose Expansion Cohorts | Up to approximately 48 months
  Overall survival is defined as the date from start of the study treatment to the date of death due to any cause.

SECONDARY OUTCOMES:
Observed Plasma Concentration of NGM707 (Including Cmax) | Baseline up to approximately 24 months
  Will be measured on Day 1, 2, 4, 8 and 15 of Cycles 1 and 3, Day 1 of Cycle 2 and Day 1 of Cycle 4 and each cycle thereafter.
Area Under the Curve (AUC) of Plasma NGM707 | Baseline up to approximately 24 months
  Area under the curve from time zero extrapolated to the last quantifiable dose of NGM707. Time zero extrapolated to the last quantifiable time point prior to the next dose. Will be measured on Day 1, 2, 4, 8 and 15 of Cycles 1 and 3, Day 1 of Cycle 2 and Day 1 of Cycle 4 and each cycle thereafter.
Plasma Half-life (t1/2) of NGM707 | Baseline up to approximately 24 months
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half. Will be measured on Day 1, 2, 4, 8 and 15 of Cycles 1 and 3, Day 1 of Cycle 2 and Day 1 of Cycle 4 and each cycle thereafter.
Anti-drug Antibodies (ADA) Against NGM707 | Baseline up to approximately 24 months
  Incidence and titers of anti-drug antibodies (ADA) against NGM707. Will be measured on Day 1 of each cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — NGM Biopharmaceuticals, Inc
Locations (23):
- United States (18):
  - NGM Clinical Study Site, Los Angeles, California
  - NGM Clinical Study Site, Newport Beach, California
  - NGM Clinical Study Site, Santa Monica, California
  - NGM Clinical Study Site, Santa Rosa, California
  - NGM Clinical Study Site, Lone Tree, Colorado
  - NGM Clinical Study Site, Washington D.C., District of Columbia
  - NGM Clinical Study Site, Sarasota, Florida
  - NGM Clinical Study Site, Baltimore, Maryland
  - NGM Clinical Study Site, Boston, Massachusetts
  - NGM Clinical Study Site, Grand Rapids, Michigan
  - NGM Clinical Study Site, Omaha, Nebraska
  - NGM Clinical Study Site, Albany, New York
  - NGM Clinical Study Site, Greenville, South Carolina
  - NGM Clinical Study Site, Dallas, Texas
  - NGM Clinical Study Site, Houston, Texas
  - NGM Clinical Study Site, San Antonio, Texas
  - NGM Clinical Study Site, Blacksburg, Virginia
  - NGM Clinical Study Site, Vancouver, Washington
- NGM Clinical Study Site, Seoul, South Korea
- Taiwan (4):
  - NGM Clinical Study Site, New Taipei City
  - NGM Clinical Study Site, Taichung
  - NGM Clinical Study Site, Tainan
  - NGM Clinical Study Site, Taipei